CLINICAL TRIAL: NCT06078501
Title: Misoprostol Effect on Second Trimester Abortion Blood Loss
Acronym: MORESTABL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment not feasible for this patient population within study timeframe
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 72229
Record Dates: First submitted 2023-10-05; First posted 2023-10-12 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Blood Loss, Surgical; Second Trimester Abortion
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misoprostol 400mcg buccal (Experimental): Participants will take 400mcg buccal misoprostol 2-3 hours prior to their procedure
  Interventions: Drug: Misoprostol 400mcg buccal
- Placebo (Placebo Comparator): Participants will take a placebo buccally 2-3 hours prior to their procedure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol 400mcg buccal — Misoprostol 400mcg buccal administration 2-3 hours prior to procedure
  Other Names: cytotec
  Arms: Misoprostol 400mcg buccal
Drug: Placebo — Placebo buccal administration 2-3 hours prior to procedure
  Arms: Placebo

SUMMARY:
Although serious complications from second trimester abortion are rare hemorrhage is the most common cause of procedural abortion related morbidity and mortality. Misoprostol is a prostaglandin E1 analogue that is used by 75% of clinicians prior to procedural abortion for the purpose of cervical preparation. Misoprostol is also known to decrease blood loss in first trimester abortion and is used to treat postpartum hemorrhage, however the effect of preprocedural misoprostol on procedural blood loss is not well described.

We will conduct a double blinded placebo-controlled gestational age stratified superiority trial of those undergoing procedural abortion between 18 and 23 weeks gestation at Stanford Health care. Participants will be randomized to either 400mcg buccal misoprostol or placebo on the day of the procedure. A quantified blood loss (QBL) will be measured during the procedure and participants will complete a survey to assess symptoms. Our primary outcome is quantified blood loss. Secondary outcomes include clinical interventions to manage excess bleeding, total procedure time, provider reported experience, patient reported experience.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant people, 18 years of age or older; intrauterine pregnancy between 18/0-23/6 weeks of gestational age (by ultrasound dating performed prior to same day of enrollment visit) consented for an induced abortion; English or Spanish speaking, able to consent for a research study, literate in English or Spanish.

Exclusion Criteria:

* known coagulopathy, suspected morbidly adherent placenta spectrum, multiple gestation, current infection, ruptured membranes, or fetal demise at time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Misoprostol 400mcg Buccal: Participants take 400mcg buccal misoprostol 2-3 hours prior to their procedure
- Placebo: Participants take a placebo buccally 2-3 hours prior to their procedure
Period: Overall Study
Arm/Group | Misoprostol 400mcg Buccal | Placebo
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Misoprostol 400mcg Buccal | Placebo | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 0 | 2
  Black or African American | 0 | 2 | 2
  Indian | 1 | 0 | 1
  Chinese | 0 | 1 | 1
  Mexican | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hemorrhage Greater Than 500 mL as a Measure of Quantified Blood Loss
Description: Quantified blood loss calculated using a combination of gravimetric and direct measurements of drapes, suction contents, and suction container.
Time Frame: day of procedure (approximately 1 hour)
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol 400mcg Buccal | Placebo
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

2. Secondary Outcome: Patient-reported Pain Scale Score
Description: Pain rated on a scale of 0 (no pain) to 10 (worst pain imaginable).
Time Frame: Day of procedure: before medication administration (2-3 hours prior to procedure); and after medication administration (up to 1 hour following completion of procedure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Misoprostol 400mcg Buccal | Placebo
Number analyzed (Participants) | 4 | 3
score on a scale
  Before medication administration | 5.00 (2.45) | 4.00 (3.46)
  After medication administration | 4.50 (4.95) | 4.00 (3.46)
Statistical Analysis 1: Comparison: Misoprostol 400mcg Buccal vs Placebo; Test type: Other; p = 0.695, Mann-Whitney U test — The a priori threshold for statistical significance was <0.05

3. Secondary Outcome: Overall Satisfaction With Care Experience Scale Score
Description: Satisfaction rated on a scale of 0 (not satisfied) to 10 (most satisfied).
Time Frame: after procedure (approximately 1 minute to complete survey)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Misoprostol 400mcg Buccal | Placebo
Number analyzed (Participants) | 4 | 3
score on a scale | 10 (0) | 10 (0)
Statistical Analysis 1: Comparison: Misoprostol 400mcg Buccal vs Placebo; Test type: Other; p = 0.91, Mann-Whitney U test; The a priori threshold for statistical significance was <0.05

4. Secondary Outcome: Number of Participants With Vaginal Bleeding
Description: Vaginal bleeding is an anticipated part of the procedure and is not always considered to be an adverse event.
Time Frame: during procedure (up to 1 hour), after medication administration
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol 400mcg Buccal | Placebo
Number analyzed (Participants) | 4 | 3
Participants | 3 | 2
Statistical Analysis 1: Comparison: Misoprostol 400mcg Buccal vs Placebo; Test type: Other; p = 1.0, Fisher Exact — The a priori threshold for statistical significance was <0.05

5. Secondary Outcome: Number of Participants With Abdominal Pain
Description: Abdominal pain is an anticipated part of the procedure and is not always considered to be an adverse event.
Time Frame: during procedure (up to 1 hour), after medication administration
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol 400mcg Buccal | Placebo
Number analyzed (Participants) | 4 | 3
Participants | 2 | 1
Statistical Analysis 1: Comparison: Misoprostol 400mcg Buccal vs Placebo; Test type: Other; p = 1.0, Fisher Exact — The a priori threshold for statistical significance was <0.05

6. Secondary Outcome: Procedure Time
Time Frame: up to 1 hour
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Misoprostol 400mcg Buccal | Placebo
Number analyzed (Participants) | 4 | 3
minutes | 22.25 (14.38) | 24.00 (15.72)
Statistical Analysis 1: Comparison: Misoprostol 400mcg Buccal vs Placebo; Test type: Other; p = 0.887, Mann-Whitney U test — The a priori threshold for statistical significance was <0.05

7. Secondary Outcome: Physician-rated Ease of Use Scale Score
Description: Ease of use rated from 1 (easiest) to 10 (most difficult)
Time Frame: after procedure (approximately 1 minute to complete survey)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Misoprostol 400mcg Buccal | Placebo
Number analyzed (Participants) | 4 | 3
score on a scale | 4.50 [3.25 to 5.75] | 5.50 [4.75 to 6.25]
Statistical Analysis 1: Comparison: Misoprostol 400mcg Buccal vs Placebo; Test type: Other; p = 0.887, Mann-Whitney U test — The a priori threshold for statistical significance was <0.05

8. Secondary Outcome: Number of Participants Estimated Blood Loss >500 ml
Description: Estimated Blood Loss calculated by subjective visual estimate based on visible blood on instruments, drapes, and suction container contents.
Time Frame: during procedure (up to 1 hour)
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol 400mcg Buccal | Placebo
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

9. Secondary Outcome: Number of Participants Requiring Manual Dilation
Time Frame: during procedure (up to 1 hour)
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol 400mcg Buccal | Placebo
Number analyzed (Participants) | 4 | 3
Participants | 1 | 1
Statistical Analysis 1: Comparison: Misoprostol 400mcg Buccal vs Placebo; Test type: Other; p = 1.0, Fisher Exact

10. Secondary Outcome: Physician-rated Satisfaction With Dilation Scale Score
Description: Satisfaction rated from 1 (least satisfied) to 10 (most satisfied)
Time Frame: after procedure (approximately 1 minute to complete survey)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Misoprostol 400mcg Buccal | Placebo
Number analyzed (Participants) | 4 | 3
score on a scale | 6.50 [5.25 to 7.75] | 8.00 [8.00 to 8.00]
Statistical Analysis 1: Comparison: Misoprostol 400mcg Buccal vs Placebo; Test type: Other; p = 1.0, Mann-Whitney U test — The a priori threshold for statistical significance was <0.05

11. Secondary Outcome: Clinician Correctly Guessed Group to Which Participant Was Randomized
Time Frame: after procedure (approximately 1 minute to complete survey)
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol 400mcg Buccal | Placebo
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0
Statistical Analysis 1: Comparison: Misoprostol 400mcg Buccal vs Placebo; Test type: Other; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Misoprostol 400mcg Buccal | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Misoprostol 400mcg Buccal (N=4) | Placebo (N=3)
Cramping (Reproductive system and breast disorders) | 4 (9) | 3 (5)

LIMITATIONS AND CAVEATS:
Early termination led to a small number of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT06078501/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT06078501/SAP_001.pdf